CLINICAL TRIAL: NCT00563017
Title: Evaluation of Efficacy and Safety of Long-acting Risperidone Microspheres in Patients With Schizophrenia or Other Psychotic Disorders When Switching From Typical Antipsychotic (Oral/Depot) or Atypical Oral Other Than Risperidone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: KW / EX / 04 - 038; HARECCTR0500047
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia, Catatonic; Schizophrenia, Disorganized; Schizophrenia, Paranoid; Schizophrenia; Psychotic Disorders
Keywords: Catatonic Schizophrenia; Disorganized Schizophrenia; Paranoid Schizophrenia; Undifferentiated Schizophrenia; Schizo-affective disorders
MeSH Terms: conditions — Schizophrenia, Catatonic; Schizophrenia, Disorganized; Schizophrenia, Paranoid; Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: Long-acting Risperidone microspheres injection

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and safety of patients on long-acting Risperidone microshpheres injection. The major advantage of long-acting injection over oral medication is facilitation of compliance in medication taking. Non-compliance is very common among schizophrenic and is a frequent cause of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with schizophrenia or another psychotic disorder according to DSM IV criteria who requires long term antipsychotic therapy
* Currently treated with either an atypical antipsychotic, other than risperidone, a conventional depot antipsychotic or oral conventional antipsychotic
* Subject has been symptomatically stable on a stable dose of an antipsychotic the last month
* Subject and/or patient's relative, guardian or legal representative has signed the informed consent form

Exclusion Criteria:

* First antipsychotic treatment ever
* On clozapine during the last 3 month
* Serious unstable medical condition
* History or current symptoms of tardive dyskinesia
* History of neuroleptic malignant syndrome
* Pregnant or breast-feeding female
* Female patient of childbearing potential without adequate contraception.
* Participation in an investigational drug trial in the 30 days prior to selection
* Known intolerance/non-responder to risperidone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-10; Study Completion 2005-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy/ Clinical Global Impression | Week 0, 4, 8,12
Personal and Social Performance Scale | Week 0, 12
Extrapyramidal Symptom | Week 0, 4, 8,12

SECONDARY OUTCOMES:
+Quality of life SF-36 | Week 0,12
Pain assoicated with injection VAS | Week 0, 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Wing King Lee, Dr, Principal Investigator — Yaumatei Psychiatric Center, Kwai Chung Hospital
Locations (1):
- Kwai Chung Hospital, Hong Kong, China